CLINICAL TRIAL: NCT04024059
Title: Contingency Management to Enhance Office-Based Buprenorphine Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00220692
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Buprenorphine Adherence and Opiate Abstinence (Experimental): Participants will receive financial incentives for buprenorphine use and opiate abstinence.
  Interventions: Behavioral: Contingency Management for adherence; Behavioral: Contingency Management for abstinence
- Buprenorphine Adherence Only (Experimental): Participants will receive financial incentives for buprenorphine use.
  Interventions: Behavioral: Contingency Management for adherence
- Control (No Intervention): Participants will not receive any intervention.

INTERVENTIONS:
Behavioral: Contingency Management for adherence — Incentives contingent on buprenorphine adherence
  Arms: Buprenorphine Adherence Only; Buprenorphine Adherence and Opiate Abstinence
Behavioral: Contingency Management for abstinence — Incentives contingent on opiate abstinence
  Arms: Buprenorphine Adherence and Opiate Abstinence

SUMMARY:
Contingency Management interventions provide incentives to substance abuse patients when patients meet therapeutic goals. This project will compare the effectiveness of two Contingency Management interventions (which the investigators have named "Buprenorphine Adherence and Opiate Abstinence" and "Buprenorphine Adherence Only") and Standard Medical Management for treating adults with opioid use disorder. Participants (N=375) will be randomly assigned to one of the three groups. Buprenorphine Adherence and Opiate Abstinence and Buprenorphine Adherence Only participants will receive incentives for daily buprenorphine use. Buprenorphine Adherence and Opiate Abstinence participants also will receive incentives for providing opiate-negative saliva samples. Daily buprenorphine use and opiate abstinence will both be remotely verified using smartphone-enabled video directly observed therapy (Video DOT). All participants will be receiving or referred to receive buprenorphine treatment and will complete assessments every 4 weeks during a 12-week intervention period.

DETAILED DESCRIPTION:
Opioid use has increased to epidemic levels in the United States and has been associated with a dramatic increase in overdose deaths. Buprenorphine is a safe, well-tolerated, and evidence-based medication for opioid use disorder that can be prescribed in office-based treatment settings. Office-based buprenorphine could be an effective way to expand treatment for opioid use disorder, and thereby combat the opioid epidemic. However, office-based buprenorphine has three limitations that must be addressed to facilitate the safe and effective expansion of buprenorphine treatment: 1) Many patients discontinue buprenorphine treatment prematurely, 2) some patients divert buprenorphine for illicit use, and 3) many patients continue to use illicit opioids during buprenorphine treatment. This project will address these limitations by using a psychosocial approach known as Contingency Management. Contingency Management interventions provide incentives to substance abuse patients when patients meet therapeutic goals. This project will compare the effectiveness of two Contingency Management interventions (which the investigators have named "Buprenorphine Adherence and Opiate Abstinence" and "Buprenorphine Adherence Only") and Standard Medical Management for treating adults with opioid use disorder. Participants (N=375) will be randomly assigned to one of the three groups. Buprenorphine Adherence and Opiate Abstinence and Buprenorphine Adherence Only participants will receive incentives for daily buprenorphine use. Buprenorphine Adherence and Opiate Abstinence participants also will receive incentives for providing opiate-negative saliva samples. Daily buprenorphine use and opiate abstinence will both be remotely verified using smartphone-enabled video directly observed therapy (Video DOT). All participants will be receiving or referred to receive buprenorphine treatment and will complete assessments every 4 weeks during a 12-week intervention period. If the proposed intervention is effective, it could encourage medical professionals to prescribe buprenorphine, and improve patients' access to and success in office-based buprenorphine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Opioid use disorder
* Enrolled in buprenorphine treatment

Exclusion Criteria:

* Unwilling or unable to use a smartphone

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Silverman, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Center for Learning and Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buprenorphine Adherence and Opiate Abstinence | Buprenorphine Adherence Only | Control
Started | 123 | 128 | 124
Completed | 112 | 126 | 119
Not Completed | 11 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine Adherence and Opiate Abstinence | Buprenorphine Adherence Only | Control | Total
Number analyzed (Participants) | 123 | 128 | 124 | 375
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 119 | 127 | 124 | 370
  >=65 years | 4 | 1 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (11) | 42 (10) | 41 (10) | 42 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 62 | 48 | 151
  Male | 82 | 66 | 76 | 224
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 4 | 7
  Not Hispanic or Latino | 122 | 126 | 120 | 368
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 3 | 7
  Asian | 3 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 36 | 24 | 33 | 93
  White | 82 | 97 | 84 | 263
  More than one race | 0 | 3 | 2 | 5
  Unknown or Not Reported | 1 | 1 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 123 | 128 | 124 | 375

OUTCOME MEASURES:

1. Primary Outcome: Buprenorphine Adherence as Assessed by the Percentage of Buprenorphine-positive Urine Samples
Description: This will be assessed by the percentage of buprenorphine-positive urine samples during the 12-week intervention.
Time Frame: 12 weeks
Measure: Number; unit: percentage of urine samples
Units Other Than Participants: urine samples
Arm/Group | Buprenorphine Adherence and Opiate Abstinence | Buprenorphine Adherence Only | Control
Number analyzed (Participants) | 123 | 128 | 124
Number analyzed (urine samples) | 369 | 384 | 372
percentage of urine samples | 80 | 84 | 78
Statistical Analysis 1: Comparison: Buprenorphine Adherence Only vs Control; Test type: Superiority; p = 0.22, Regression, Logistic; Odds Ratio (OR) = 1.737, 95% CI 2-sided [0.719 to 4.195]
Statistical Analysis 2: Comparison: Buprenorphine Adherence and Opiate Abstinence vs Control; Test type: Superiority; p = 0.938, Regression, Logistic; Odds Ratio (OR) = 1.035, 95% CI 2-sided [0.435 to 2.461]

2. Primary Outcome: Opiate Abstinence as Assessed by the Percentage of Opiate-negative Urine Samples
Description: This will be assessed by the percentage of opiate-negative urine samples during the 12-week intervention.
Time Frame: 12 weeks
Measure: Number; unit: percentage of urine samples
Units Other Than Participants: urine samples
Arm/Group | Buprenorphine Adherence and Opiate Abstinence | Buprenorphine Adherence Only | Control
Number analyzed (Participants) | 123 | 128 | 124
Number analyzed (urine samples) | 369 | 384 | 372
percentage of urine samples | 83 | 85 | 80
Statistical Analysis 1: Comparison: Buprenorphine Adherence Only vs Control; Test type: Superiority; p = 0.202, Regression, Logistic; Odds Ratio (OR) = 1.783, 95% CI 2-sided [0.733 to 4.336]
Statistical Analysis 2: Comparison: Buprenorphine Adherence and Opiate Abstinence vs Control; Test type: Superiority; p = .474, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.571 to 3.336]

3. Secondary Outcome: Buprenorphine Diversion as Assessed by Percentage of Participants Reporting Any Diversion of Buprenorphine
Description: This is the percentage of participants reporting any diversion of buprenorphine at each assessment during the 12-week intervention.
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Buprenorphine Adherence and Opiate Abstinence | Buprenorphine Adherence Only | Control
Number analyzed (Participants) | 123 | 128 | 124
percentage of participants | 16.12 | 16.28 | 18.82
Statistical Analysis 1: Comparison: Buprenorphine Adherence Only vs Control; Test type: Superiority; p = 0.328, Regression, Logistic; Odds Ratio (OR) = 0.669, 95% CI 2-sided [0.299 to 1.497]
Statistical Analysis 2: Comparison: Buprenorphine Adherence and Opiate Abstinence vs Control; Test type: Superiority; p = 0.435, Regression, Logistic; Odds Ratio (OR) = 0.724, 95% CI 2-sided [0.322 to 1.627]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Buprenorphine Adherence and Opiate Abstinence | Buprenorphine Adherence Only | Control
All-Cause Mortality (participants affected / at risk) | 1/123 | 0/128 | 0/124
Serious Adverse Events (participants affected / at risk) | 5/123 | 4/128 | 2/124
Other Adverse Events (participants affected / at risk) | 0/123 | 0/128 | 0/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine Adherence and Opiate Abstinence (N=123) | Buprenorphine Adherence Only (N=128) | Control (N=124)
Breast Cancer (General disorders) | 0 (0) | 1 (1) | 0 (0)
Assault (General disorders) | 0 (0) | 1 (1) | 0 (0)
Covid (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
endocarditis with heart surgery for pace maker (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Psychiatric (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
blood clot in lungs (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT04024059/Prot_SAP_000.pdf